CLINICAL TRIAL: NCT07152717
Title: Assessment of a Connected-health, Pressure Monitoring Technology for Improving Clinical Outcomes of Compression Therapy in the Treatment of Venous Leg Ulcers
Brief Title: Assessing Connected-Health, Pressure-Monitoring Technology for Improving Compression Therapy in Venous Leg Ulcer Treatment
Acronym: ACHIEVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Feeltect Limited (Industry)
Collaborators: Parkview Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUR25-0409WoundCompress
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Venous Leg Ulcers (VLUs)
Keywords: wound care; compression therapy; venous leg ulcers; remote monitoring; pressure sensing; connected health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Cohort (Other): Patients will receive their normal standard of care and usual pattern of wound care visits from the treating provider. The Tight Alright device will be placed under the compression wrap by a study investigator and data will be transmitted but blinded to clinicians and patients. All patients in the Control Cohort will complete the study prior to initiating patients into the Intervention Cohort.
  Interventions: Device: A connected-health, pressure-sensing system for monitoring sub-bandage pressure during compression therapy
- Intervention Cohort (Experimental): Patients will receive their normal standard of care with the addition of using the Tight Alright technology, applied by a study investigator, to guide the application of compression to targeted pressures. The Tight Alright technology will be used to monitor pressure in the home setting, using the app (point-of-care) and web-dashboard (remotely), and to guide the reapplication of targeted pressure. If pressures drop below 40 mmHg at the B sensor, for two consecutive readings, reapplications will be considered. Reapplication of compression using a top-up layer can be delivered in a number of different ways, including additional patient visits, patient, informal caregiver, self-management via teleconsultation, or independent self-management.
  Interventions: Device: A connected-health, pressure-sensing system for monitoring sub-bandage pressure during compression therapy

INTERVENTIONS:
Device: A connected-health, pressure-sensing system for monitoring sub-bandage pressure during compression therapy — The Tight Alright system, developed by FeelTect Limited, consists of a wearable, pressure sensing device that measures sub-bandage pressure at three regions along the length of the lower leg. The wearable device transmits data wirelessly to a mobile app on a smart device, which then displays the data in real-time. The mobile app is also capable of transmitting data to a remote cloud database, via the internet, where it can be viewed on a remote dashboard (i.e., via a secure webpage).
  Other Names: FeelTect Tight Alright

SUMMARY:
This study evaluates the effectiveness of a connected-health, pressure monitoring technology (Tight Alright) to improve clinical outcomes of compression therapy in patients with venous leg ulcers (VLUs). Compression therapy is the standard of care for VLUs, but achieving and maintaining therapeutic sub-bandage pressure is challenging due to patient variability and lack of objective feedback. The Tight Alright system includes a wearable device that measures sub-bandage pressure at multiple points on the leg and transmits data to a mobile app and cloud database, enabling both guided compression application at the point-of-care and guided compression maintenance via remote monitoring.

The study will be conducted at Parkview Noble Center for Wound Healing and will include two cohorts: a control group receiving standard unguided compression therapy with blinded device use (i.e. compression pressures will be blinded at the point of care but monitored remotely), and an intervention group using Tight Alright technology to guide compression application and reapplication. Outcomes will include wound healing rates, time to healing, pressure maintenance, patient adherence, and usability. The study aims to determine whether integrating connected-health pressure monitoring can improve consistency of compression therapy, accelerate healing, and enhance patient engagement in the treatment of venous leg ulcers

ELIGIBILITY:
Inclusion Criteria:

* Patient of Parkview Noble Center for Wound Healing
* Adults 18+ with venous leg ulcers receiving compression therapy treatment prescribed by outpatient wound clinic.
* Capable of using use a smart device
* Owns a smart phone or device capable of downloading the Mobile App

Exclusion Criteria:

* <18 years old
* Unable to consent in English
* Cellulitis in affected limb
* Acute deep vein thrombosis in affected limb
* Active malignancy in affected limb
* Prisoners
* Currently enrolled in or has been enrolled in another investigation device or drug trial in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage area reduction per day | From enrollment to the end of treatment at 5 weeks
  The daily rate of wound area reduction represented as a percentage, calculated by comparing the wound size at the end of the treatment (Aend) with the wound size at the start of treatment (Astart) and normalising for the length of time for treatment (T). (Aend - Astart)/Astart*100/T

SECONDARY OUTCOMES:
Average pressure | From enrollment to the end of treatment at 5 weeks
  The average pressure applied over the duration of treatment
Percentage of patients healed | From enrollment to the end of treatment at 5 weeks
  The percentage of patients healed completely within the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Parkview Center for Wound Healing, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 1 month and ending 3 years after the publication of results
Access Criteria: IPD will be shared if there is a legitimate concern, as assessed by the clinical team executing the study in Parkview Health, raised by other researchers about the validity of the data or the data processing methods, including statistical analysis. Brooke Randol will make the final decision on sharing IPD. An appropriate mechanism will be negotiated for sharing data, which may include a request for the proposed data analysis by other researchers and a data sharing agreement.